CLINICAL TRIAL: NCT06562920
Title: A Single-arm, Prospective, Exploratory Study of Adebrelimab Combined With Chemotherapy and Concurrent SBRT for Neoadjuvant Treatment of Limited-stage Small Cell Lung Cancer and Analysis of Biological Markers（ASSESS）
Brief Title: Adebrelimab Combined With Chemotherapy and Concurrent SBRT for Neoadjuvant Treatment of Limited-stage Small Cell Lung Cancer
Acronym: Neoadjuvant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, liujinshi, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-738 (IIT)
Record Dates: First submitted 2024-08-06; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Efficacy and Safety of Neoadjuvant Immunotherapy for Small Cell Lung Cancer
Keywords: small cell lung cancer; Neoadjuvant immunotherapy; SBRT
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This study plans to enroll 20 patients with previously untreated T1-3N0-1M0 resectable limited-stage small cell lung cancer. They will receive 3 cycles of adebrelimab combined with chemotherapy and concurrent SBRT, and undergo surgery within 4-6 weeks after treatment. After surgery, adjuvant therapy will be considered based on the results of MDT discussion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant anti-PDL-1 Immunotherapy combined chemotherapy and SBRT (Experimental): Three cycles of neoadjuvant PDL-1 combined chemotherapy and SBRT followed by surgery for limited-stage small cell lung cancer
  Interventions: Drug: adebrelimab and chemotherapy

INTERVENTIONS:
Drug: adebrelimab and chemotherapy — 3 cycles of adebrelimab combined with chemotherapy and concurrent SBRT, and undergo surgery within 4-6 weeks after treatment.
  Other Names: SBRT

SUMMARY:
To explore the effectiveness and safety of adebrelimab combined with chemotherapy and concurrent SBRT for 3 cycles of neoadjuvant treatment followed by surgery in T1-3N0-1M0 limited-stage SCLC

DETAILED DESCRIPTION:
This study plans to enroll 20 patients with resectable limited-stage small cell lung cancer in stage T1-3N0-1M0 who have not been treated before. They will receive 3 cycles of adebelimumab combined with chemotherapy and concurrent SBRT. Surgery will be performed within 4-6 weeks after treatment. After surgery, adjuvant therapy will be considered based on the results of MDT discussion. All patients with tumor recurrence and metastasis will enter survival follow-up. Pathological complete response rate (pCR) and safety indexes were used as the main observation indicators.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old; Histologically or cytologically confirmed as limited-stage small cell lung cancer (T1-3N0-1M0); All lesions of the patient (including primary lesions, lymph nodes/metastatic lesions assessed as metastases) must be jointly evaluated by surgeons, radiotherapists, and radiologists to be surgically resectable; Subjects must have measurable target lesions (according to RECIST 1.1 standards); ECOG performance status score 0-1; No history of other malignant tumors; No previous anti-tumor treatment such as surgery, radiotherapy, chemotherapy, immunotherapy, etc. related to small cell lung cancer; Patients must have sufficient cardiopulmonary function: FEV1 and DLCO of patients are ≥50% of the predicted value, echocardiography indicates LVEF ≥55%, and no clear signs of heart failure, severe coronary artery stenosis, etc. are found in various tests. Cardiopulmonary function is assessed by surgeons to be able to tolerate surgical treatment;

The functional level of each important organ must meet the following requirements:

1. Bone marrow: absolute neutrophil count (ANC) ≥1.5× 109/L, platelets ≥100 × 109/L, hemoglobin ≥9 g/dl;
2. Good coagulation function: defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
3. Liver: total bilirubin ≤1.5 times the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal;
4. Kidney: serum creatinine ≤1.25 times the upper limit of normal or creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min; Men of childbearing potential and women of childbearing age must agree to take effective contraceptive measures from the signing of the main informed consent until 180 days after the last dose of the study drug. Women of childbearing age include premenopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test result within ≤ 7 days before the first administration of the study drug; Voluntarily participate in the clinical study; fully understand and be informed of this study and sign the ICF (Informed Consent Form).

Exclusion Criteria:

* All lesions cannot be completely removed by surgery. Received anti-tumor treatment for SCLC (including but not limited to chemotherapy, radiotherapy of the lesion site); Previously used immune checkpoint inhibitors such as PD-1/PD-L1 inhibitors; Any active autoimmune disease or history of autoimmune disease (such as uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after hormone replacement therapy), tuberculosis); Patients with complete remission of childhood asthma and no need for any intervention as an adult or vitiligo can be included, but patients who require bronchodilators for medical intervention are not included; Suffering from congenital or acquired immune deficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method) or co-infection with hepatitis B and hepatitis C; Presence of difficult-to-control third-cavity effusion, such as large pleural effusion or ascites or pericardial effusion; Presence of huge mediastinal masses, multiple lesions, extracapsular invasion or fusion of complex small cell lung cancer; Subjects who need systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressants within 14 days before the first medication. In the absence of active autoimmune diseases, inhaled or topical corticosteroids and adrenal hormone replacement therapy with a dose of >10 mg/day of prednisone at an effective dose are allowed; Subjects who have been treated with anti-tumor vaccines or other anti-tumor drugs with immunostimulatory effects (interferon, interleukin, thymosin, immune cell therapy, etc.) within 1 month before the first medication; Subjects who are participating in other clinical studies or whose first medication time is less than 4 weeks (or 5 half-lives of the study drug) from the end of the previous clinical study (last dose); Evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, and severe lung function impairment, etc.; Combined with severe heart disease Patients with congestive heart failure of grade III or above (NYHA standard), or angina of grade III or above (CCS standard), or a history of myocardial infarction within 6 months before the start of treatment, or arrhythmia requiring drug treatment; Major surgery, open biopsy or significant trauma within 28 days before enrollment; A known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; Pregnant or lactating women; patients of childbearing potential who are unwilling or unable to take effective contraceptive measures; Known to have allergic reactions, hypersensitivity reactions or intolerance to study drugs Other conditions that the investigator believes are not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
pCR | Assessed average of 1 month after surgery
  Pathological Complete Response
Safety and Tolerability | Assessed average of 1 month after surgery
  Adverse reactions (according to CTCAE v5 classification)

SECONDARY OUTCOMES:
MPR | Assessed average of 1 month after surgery
  Major Pathological response
Event-Free Survival(EFS) | From the time of enrollment, until the disease relapses or metastasizes，assessed up to 5 years follow-up.
  Refers to the time from randomization to the first occurrence of any of the following events: disease progression that is inoperable, local or distant recurrence, death due to any cause, etc.
Objective Response Rate(ORR) | From the time of enrollment, assessed before surgery
  The proportion of patients whose tumors shrink to a certain amount and remain shrinking for a certain period of time includes complete remission (CR) and partial remission (PR).
Overall survival(OS) | From the time of enrollment, assessed up to 5 years follow-up.
  The time from the start of treatment to the death of the subject due to various causes was calculated based on the intention-to-treat population (ITT).
Exploration of tumor efficacy markers | From the time of enrollment, assessed up to 5 years follow-up.
  Correlation between MRD biomarkers in tumor tissue and peripheral blood and patients' clinical outcomes, progression, and efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No